CLINICAL TRIAL: NCT05661838
Title: Effect of Intraoperative Allogeneic Blood Transfusion on Postoperative Pulmonary Complications in Elective Spinal Surgery: a Retrospective Cohort Study
Brief Title: Effect of Intraoperative Allogeneic Blood Transfusion on Postoperative Pulmonary Complications
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-0968
Record Dates: First submitted 2022-12-15; First posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2013-08

CONDITIONS: Spinal Fusion; Transfusion; Pulmonary Complication
MeSH Terms: interventions — Blood Transfusion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- non-PPCs group: Patients without PPCs (Pleural effusion, Pulmonary atelectasis, Pulmonary infection)
  Interventions: Procedure: transfusion
- PPCs group: Patients with PPCs (Pleural effusion, Pulmonary atelectasis, Pulmonary infection)
  Interventions: Procedure: transfusion

INTERVENTIONS:
Procedure: transfusion — transfusion

SUMMARY:
Elective spine surgery is associated with a high incidence of perioperative complications, including peri- and postoperative pulmonary complications (PPCs), which occur in nearly 4% of patients. More than 40% of all deaths after elective spine surgery are attributed to PPCs. However, whether it influences risk of other PPCs is unclear.

ELIGIBILITY:
Inclusion Criteria:

* Patients were included if they underwent elective spine surgery (e.g. multi-segmental thoracic, lumbar, or thoracolumbar spine surgery) at the Second Hospital of Zhejiang University School of Medicine from August 1, 2013 to October 31, 2020

Exclusion Criteria:

* combined anterior-posterior surgery
* growth rod adjustment surgery
* spinal tumor.
* surgery took fewer than 3 hours.

Ages: 9 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients were included if they underwent post vertebral column resection (e.g. multi-segmental thoracic, lumbar, or thoracolumbar spine surgery) at the Second Hospital of Zhejiang University School of Medicine from August 1, 2013 to October 31, 2020
Sampling Method: Probability Sample
Enrollment: 272 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Correlation between blood transfusion and postoperative pulmonary complications | 28 days after surgery
  Correlation between blood transfusion and postoperative pulmonary complications

CONTACTS AND LOCATIONS:
Overall Officials: Min Yan, doctor, Study Chair — The Second Affiliated Hospital of Zhejiang University Medical College
Locations (1):
- The Second Affiliated Hospital of Zhejiang University anesthesiology department, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided